CLINICAL TRIAL: NCT03281993
Title: Alternative Apnea Test as the Method of Brain Death Diagnosis .
Brief Title: Apnea Tests as the Methods of Brain Death Diagnosis.
Acronym: DiagBD
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Joanna Sołek-Pastuszka, MD PhD, Pomeranian Medical University Szczecin
Other Study IDs: KB-0012/116/13
Record Dates: First submitted 2017-09-03; First posted 2017-09-13 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Brain Death; Apnea; Pupillary Anomaly
Keywords: apnea test, brain death, pupillometry
MeSH Terms: conditions — Brain Death; Apnea; Pupil Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CPAP-AT: After 2 hours from I-AT was performed the alternative AT by CPAP ventilation mode. Before CPAP-AT and 10 minutes after blood samples for arterial blood gases (ABG) were collected. If the investigators observe rapid desaturation defined as a decline in O2 saturation below 85%, CPAP-AT was aborterd.
  Interventions: Other: CPAP AT

INTERVENTIONS:
Other: CPAP AT — If the investigators observe rapid desaturation defined as a decline in O2 saturation below 85%; the CPAP apnea test (CPAP-AT) test was aborted.
  Other Names: change type of ventylation

SUMMARY:
Apnea test (AT) is the most important clinical test performed usually at the end of brain death (BD) diagnosis procedure. Traditional insufflation apnea test (I-AT) cannot be completed in patients with extremely compromised lung function due to rapid blood desaturation and circulatory disturbances. Therefore the investigators decided to verify alternative AT options such as continuous positive airway pressure apnea test (CPAP-AT) in patients with good and poor baseline oxygenation, before implementing them in currently reviewed Polish BD criteria.

DETAILED DESCRIPTION:
Apnea test (AT) is one of the most important examination during the diagnosis of brain death. It is usually performed at the end of each series of clinical examinations during diagnostic process. The most popular standard insufflation apnea test (I-AT) may be potentially harmful. It may cause some serious complications including pneumothorax, severe hypoxemia, hemodynamic instability and even cardiac arrest. Therefore, the investigators decided to analyze apnea test in CPAP option (CPAP-AT) as a new tool. For safety of the study the investigators analyzed a method after BD diagnosis.

Methods:

I-AT and hypoventilation with 100 % oxygen (if needed) were performed according to Polish guidelines. Two hours after BD diagnosis was performed extra apnea test in CPAP option (CPAP-AT). Before CPAP-AT the patients were ventilated 100% oxygen. After then the ventilator settings were changed to CPAP mode with PEEP 10 cm H2O, PS 0 cm H2O, FiO2 1,0, flow 6L/min. Emergency apnea ventilation was turned off. At the beginning of CPAP mode and 10 minutes after, blood samples for arterial blood gases (ABG) were collected. If were observed rapid desaturation defined as a decline in O2 saturation below 85%, CPAP-AT was aborted and study was finished.

During routine diagnosis of brain death, pupillary dilation after a neck flexion was observed in one case. Therefore, the investigators decided to use a pupillometer during brain death examination to find out how pupils react after a neck flexion and how often it happens.

Pupil measurements were taken immediately after the diagnosis of brain death. The measurements of pupil diameter were taken twice: A - before neck flexion; B - after neck flexion. We used pupillometer: AlgiScan (Equip Medkey BV).

ELIGIBILITY:
Inclusion Criteria:

* brain death diagnosis

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated adult ICU patients at the Intensive Care Unit of the Department of Anaesthesia and Intensive Care teaching hospital at the Pomeranian Medical University in Szczecin during Brain Death diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2015-06-25 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline arterial blood gases (ABG) during CPAP-AT | 10 minutes
  After 2 hours from I-AT was performed the alternative AT by CPAP ventilation mode. Before CPAP-AT the patients were ventilated 100% oxygen. After then the ventilator parameters were modified to: 0 H2O of pressure support (PS), 10 cm H2O of PEEP, 6l/min of O2 flow and 0.2 l/min of sensitivity. Before the test and 10 minutes after then was taken blood probe to ABG and type of ventilation change to pretest settings. The test is considered valid if there is no respiratory activity despite the rise of PaCO2 above 60mmHg and over 20mmHg above the baseline. If the investigators observe rapid desaturation defined as a decline in O2 saturation below 85%, CPAP-AT was aborterd.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Pastuszka, MD PhD, Principal Investigator — Pomeranian Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solek-Pastuszka J, Sawicki M, Iwanczuk W, Bohatyrewicz R. Ventilator-Delivered Continuous Positive Airway Pressure for Apnea Test in the Diagnosis of Brain Death in Patient With Extremely Poor Baseline Lung Function-Case Report. Transplant Proc. 2016 Sep;48(7):2471-2472. doi: 10.1016/j.transproceed.2016.02.089. PMID 27742325
- [Background] Saucha W, Solek-Pastuszka J, Bohatyrewicz R, Knapik P. Apnea test in the determination of brain death in patients treated with extracorporeal membrane oxygenation (ECMO). Anaesthesiol Intensive Ther. 2015;47(4):368-71. doi: 10.5603/AIT.2015.0051. PMID 26401745
- [Background] Solek-Pastuszka J, Saucha W, Iwanczuk W, Bohatyrewicz R. Evolution of apnoea test in brain death diagnostics. Anaesthesiol Intensive Ther. 2015;47(4):363-7. doi: 10.5603/AIT.2015.0050. PMID 26401744